CLINICAL TRIAL: NCT03779607
Title: Clinical Evaluation and Patient Satisfaction Ofshade Matching Between Natural Teeth and Monolithic All-ceramic Crowns Fabricated From Two Materials (Randomized Controlled Clinical Trial)
Brief Title: Clinical Evaluation and Patient Satisfaction of Shade Matching Between Natural Teeth and Monolithic All-ceramic Crowns Fabricated From Two Materials
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed el sayed bekhiet, Resident - Fixed prosthodontic department- Faculty of oral and dental medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-11-13
Record Dates: First submitted 2018-11-12; First posted 2018-12-19 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Natural Optical Properties

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPS e.max Press(lithium di silicate) (Active Comparator): Lithium disilicate reinforced glass ceramics are available in the market in two forms according to the technique of manufacturing, either heat pressed ingots or CAD/CAM blocks for milling. The heat pressed lithium disilicate glass ceramic consists of approximately 70% lithium disilicatecrystals(the main crystal phase) having a needle like shape that are embedded in a glassy matrix. The crystals length is about 3 to 6 μm. The heat pressed ingots are fully crystallized and the restoration is fabricated by the lost wax technique where the lithium disilicate ingots are pressed into the investment mold at high temperature. The pressed lithium disilicate has strong flexural strength values(range 400 ± 40 MPa)
  Interventions: Other: Celtra Press
- Celtra Press (Experimental): new class of zirconia-reinforced lithium silicate material available to labs for pressing. This unique material provides top aesthetics and is virtually impossible to tell apart from a natural tooth.
  Celtra Press is a multiphase ceramic consisting of a glass matrix and lithium disilicate crystals having a crystal length of about 1.5 µm plus nano-scale lithium phosphate . In addition to Li2O and SiO2, Celtra Press contains about 10% zirconia (ZrO2), which is dissolved completely in the glass phase rather than in crystalline form. Celtra Press is characterized by a high strength of about 500 MPa and excellent flow properties during pressing.
  Interventions: Other: Celtra Press

INTERVENTIONS:
Other: Celtra Press — new class of zirconia-reinforced lithium silicate material available to labs for pressing. This unique material provides top aesthetics and is virtually impossible to tell apart from a natural tooth.
  Celtra Press is a multiphase ceramic consisting of a glass matrix and lithium disilicate crystals having a crystal length of about 1.5 µm plus nano-scale lithium phosphate . In addition to Li2O and SiO2, Celtra Press contains about 10% zirconia (ZrO2), which is dissolved completely in the glass phase rather than in crystalline form. Celtra Press is characterized by a high strength of about 500 MPa and excellent flow properties during pressing.

SUMMARY:
evaluation of color difference between zirconia reinforced lithium silicate (celtra press) VS lithium disilicate (Emax) in relation to natural tooth structure to determine which monolithic material will provide restoration with exact shade and optical properties as natural tooth structure.

DETAILED DESCRIPTION:
eligible patients will be randomized in 2 equal group between study group (celtra press) and control group (Emax) .

Single tooth in esthetic zone requiring full coverage crown is prepared to receive an all ceramic crown of .

Grouping: The crowns will be divided into two groups:

I:Teeth receiving crowns fabricated from IPS emax press ( ivoclarvivadent) II:Teeth receiving crowns fabricatedfrom Celtrapress(dentsplysirona).

Shade will be measured using intraoral spectrophotometer and evaluated.

The color difference (ΔE ) will be calculated for each sample using the following equation: ΔE =[(ΔL*)²+(Δa*)² + (Δb*)²]½

ΔE (perceptibility threshold ) will be evaluated for each group.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age range of the patients from 20-45 years old; able to read and sign the informed consent document, illiterate patient will be avoided.

  2. Patients able physically and psychologically to tolerate conventional restorative procedures.

  3. Patients with no active periodontal or pulpal diseases, having teeth with good restorations.

  4. Patients with teeth problems indicated for full coverage restoration ( coronal fracture where partial coverage would lack retention, malposed or malformed teeth).

  5. Patients with root canal treated teeth requiring full coverage restorations with contralatral tooth not filled orfractured.

  6. Patients willing to return for follow-up examinations and evaluation.

Exclusion Criteria:

1. Patients in the growth stage with partially erupted teeth.
2. Patients with poor oral hygiene and motivation.
3. Pregnant women's to avoid any complication that may occur in dental office due to pregnancy or due to injected anesthetic solution.
4. Patients with psychiatric problems or unrealistic expectation
5. Patients have no opposite occluding dentition in the area intended for restoration\
6. Patients suffer from parafunctional habits.
7. deep discoloration of abutment .
8. Smokers and heavy caffeine consumers.

   -

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Color match | immediately after crown cementation
  using USPHS scoring system

SECONDARY OUTCOMES:
Patient satisfaction | immediately after crown cementation
  Patient satisfaction using Visual Analogue scale- Binary (Satisfied or not satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed zamzam, professor, Principal Investigator — Fixed Prosthodontics Faculty of Oral and dental medicine Cairo University; Maha Taymour, Associate professor, Study Director — Fixed Prosthodontics Faculty of Oral and dental medicine Cairo University

IPD SHARING:
Plan to Share IPD: Undecided